CLINICAL TRIAL: NCT02859337
Title: Improving the Effectiveness of Orally Dosed Emergency Contraceptives in Obese Women - PK and PD of 30mg and 60mg UPA
Brief Title: Effectiveness of Orally Dosed Emergency Contraception in Obese Women - UPA
Acronym: UPA-Obesity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Alison Edelman, Professor, OB/GYN, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OHSU IRB 016291
Record Dates: First submitted 2016-08-04; First posted 2016-08-09 (Estimated); Results first posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Obesity; Contraception
Keywords: obesity; body weight; BMI; emergency contraception; levonorgestrel; ulipristal acetate
MeSH Terms: conditions — Obesity; Body Weight | interventions — ulipristal acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- UPA-ECx1 followed by ECx2 (Active Comparator): Ulipristal acetate 30mg orally x 1 dose, washout cycle and then in the next menstrual cycle, 60mg x 1 dose. Timing of dosage depends on follicle measurements.
  Interventions: Drug: UPA-ECx1; Drug: UPA-ECx2
- UPA-ECx2 followed by ECx1 (Experimental): Ulipristal acetate 60mg orally x 1 dose, washout cycle, and then in next menstrual cycle 30mg orally x 1 dose. Timing of dosage depends on follicle measurements.
  Interventions: Drug: UPA-ECx1; Drug: UPA-ECx2
- UPA-ECx1 Normal BMI/weight (Other): Ulipristal acetate 30mg orally x 1 dose. timing of dosage depends on follicle measurements. This is to obtain a normal BMI control group.
  Interventions: Drug: UPA-ECx1

INTERVENTIONS:
Drug: UPA-ECx1 — Evaluating the pharmacodynamic and pharmacokinetic outcomes in obese women using 30mg of UPA-based EC
  Other Names: Ella; Ella-One
Drug: UPA-ECx2 — Evaluating the pharmacodynamic and pharmacokinetic outcomes in obese women using 60mg of UPA-based EC
  Other Names: ella; ella-one
  Arms: UPA-ECx1 followed by ECx2; UPA-ECx2 followed by ECx1

SUMMARY:
Obese women are significantly more likely than their normal BMI counterparts to experience failure of orally-dosed emergency contraceptives. Our preliminary data provides evidence for testing a dose escalation strategy in an effort to provide improved efficacy from orally-dosed emergency contraceptives in obese women. More data is needed regarding emergency contraception containing ulipristal acetate. The overall project will be focused on both levonorgestrel (LNG) - and ulipristal acetate (UPA)-containing emergency contraception but this protocol registration is for the UPA aspect of the study procedures.

DETAILED DESCRIPTION:
Emergency contraception (EC) provides a woman with an additional line of defense against unintended pregnancy following an act of unprotected intercourse. Orally-dosed EC works by delaying ovulation and reduces the risk of pregnancy for a single act of unprotected intercourse by 50-70%. Unfortunately, obese women are significantly more likely than their normal BMI counterparts to experience failure of orally-dosed EC and in some instances EC is equivalent to placebo.

Our preliminary data provides evidence for testing a dose escalation strategy in an effort to provide improved efficacy from orally-dosed EC in obese women. We hypothesize that increasing the dose of orally-dosed EC agents will normalize the pharmacokinetics resulting in the expected treatment effect (delay in follicle rupture) in obese women. In the overall proposal, we plan to perform detailed pharmacokinetic and pharmacodynamic studies of UPA-based EC in obese women and expand upon our preliminary findings of LNG-based EC. This protocol registration is for the UPA aspect of the study procedures focused on the pharmacokinetics and pharmacodynamics of UPA and will include a dose escalation intervention.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy women
* Aged 18-35 years old
* Regular menses (every 21-35 days) experiencing an ovulatory screening cycle with a progesterone level of 3 ng/mL or greater
* Subjects must have a BMI of >30kg/m2 and weight at least 80kg or more OR a BMI <25kg/m2 and a weight of less than 80kg.

Exclusion Criteria:

* Metabolic disorders including uncontrolled thyroid dysfunction and Polycystic Ovarian Syndrome
* Impaired liver or renal function
* Actively seeking or involved in a weight loss program (must be weight stable) pregnancy, breastfeeding, or seeking pregnancy
* Recent (within last 8 weeks) use of hormonal contraception
* Current use of drugs that interfere with metabolism of sex steroids
* Smokers.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2022-01-13 (Actual); Study Completion 2023-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ALISON EDELMAN, MD, MPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- OHSU, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
PI acknowledges willingness to share data and materials with other investigators through established means. Data will be shared with collaborators as soon as available; with other scientists before publication if the work to be done is different from our purposes; with local colleagues at seminars and talks including our yearly university wide research-in-progress seminar; and with the scientific community at large by posters and presentations at local, regional, national, and international scientific meetings. Data will be presented via publication to the widest audience possible.
  Transfer of resources is subject to the acceptance of a Materials Transfer Agreement as required by policy at OHSU.
  OHSU complies with NIH policy on Sharing Research Data and on Sharing Model Organisms.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | UPA-ECx1 Followed by ECx2 | UPA-ECx2 Followed by ECx1 | UPA-ECx1 Normal BMI/Weight
Started | 25 (25 completed Cycle 1 (ECx1)) | 27 (27 completed Cycle 1 (ECx2)) | 12
Completed | 19 (19 completed Cycle 3 (ECx2) and thus also completed the entire study) | 24 (24 completed Cycle 3 (ECx1) and thus also completed the entire study) | 12
Not Completed | 6 | 3 | 0
Not completed — Study drug not dosed (no dominant follicle) | 2 | 2 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Primary outcome is analyzed by cycle and dose but demographics were analyzed by group allocation
Groups:
- Total: Total of all reporting groups
Arm/Group | UPA-ECx1 Followed by ECx2 | UPA-ECx2 Followed by ECx1 | UPA-ECx1 Normal BMI/Weight | Total
Number analyzed (Participants) | 25 | 27 | 12 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (3.4) | 28.7 (3.7) | 30 (3.5) | 29.6 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 27 | 12 | 64
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Participants were able to indicate more than one Race/Ethnicity.
  Participants
    Hispanic/Latino | 2 | 5 | 0 | 7
    Not Hispanic/Latino | 23 | 22 | 12 | 57
    Asian | 1 | 0 | 2 | 3
    Black | 3 | 3 | 1 | 7
    White | 20 | 24 | 9 | 53
    Declined to specify | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 25 | 27 | 12 | 64
BMI [Mean (Standard Deviation); unit: kg/m2] | 37.9 (6.7) | 39.3 (5.4) | 22.6 (1.4) | 35.2 (8.1)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Delay in Follicular Rupture Beyond 5 Days
Description: Follicular rupture (yes/no) beyond 5 days from EC dosing by ultrasound in participants with a BMI >/=30 kg/m2. The comparison is between menstrual cycles where 30 versus 60 mg of UPA was taken. Follicular rupture is defined as the disappearance of or >50% reduction in size of the leading follicle. The day of EC dosing is defined as day zero.
Time Frame: 1 menstrual cycle, assessed up to 38 days
Population: The total analyzed number is the menstrual cycle of the participant with a BMI >/=30kg/m2 when dosed with ECx1 or ECx2 who experienced a delay in follicular rupture beyond 5 days after dosing EC.
Measure: Count of Participants; unit: Participants
Groups:
- ECx1 BMI>/=30kg/m2: Participants with a BMI >/=30kg/m2 in the cycle dosed with 30 mg UPA
- ECx2 BMI >/=30: Participants with a BMI >/=30kg/m2 in the cycle dosed with 60 mg UPA
- ECx1 BMI <25kg/m2: Control group. Participants with a BMI <25kg/m2 in the cycle dosed with 30 mg UPA.
  No planned statistical comparison analysis with the BMI >/=30 kg/m2 groups
Arm/Group | ECx1 BMI>/=30kg/m2 | ECx2 BMI >/=30 | ECx1 BMI <25kg/m2
Number analyzed (Participants) | 49 | 46 | 12
Participants | 46 | 43 | 12

2. Secondary Outcome: Maximum Serum Concentration of Ulipristal Acetate
Description: Maximum serum concentration (Cmax) of UPA in participants with BMI >/=30 kg/m2 with 30 mg UPA, with BMI >/= 30 kg/m2 with 60 mg UPA, and normal BMI participants with 30mg UPA
Time Frame: 24 hours
Population: This was a voluntary aspect of the protocol so data were only collected on a subset of the sample.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- ECx2 BMI >/=30kg/m2: Participants with a BMI >/=30kg/m2 in the cycle dosed with 60 mg UPA
- ECx1 BMI <25kg/m2: Control group. Participants with a BMI <25kg/m2 in the cycle dosed with 30 mg UPA
Arm/Group | ECx1 BMI>/=30kg/m2 | ECx2 BMI >/=30kg/m2 | ECx1 BMI <25kg/m2
Number analyzed (Participants) | 18 | 17 | 12
ng/mL | 197.1 (118.5) | 312.4 (215.3) | 98.4 (40.7)

ADVERSE EVENTS:
Time Frame: Over approximately 3 months
Description: AE/SAE are consistent with clinicaltrials.gov
Arm/Group | ECx1 BMI>/=30kg/m2 | ECx2 BMI >/=30kg/m2 | ECx1 BMI <25kg/m2
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/46 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/46 | 0/12
Other Adverse Events (participants affected / at risk) | 0/49 | 0/46 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-03-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT02859337/Prot_SAP_002.pdf
  • Informed Consent Form (2016-05-06): https://cdn.clinicaltrials.gov/large-docs/37/NCT02859337/ICF_001.pdf